CLINICAL TRIAL: NCT00076583
Title: Motor Skill Learning: Spinal Reflexes
Brief Title: Spinal Reflexes in Motor Skill Learning
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040107; 04-N-0107
Record Dates: First submitted 2004-01-26; First posted 2004-01-27 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Healthy
Keywords: Motor Learning; Co-contraction; Reciprocal Inhibition; Spinal Plasticity; Rhythmic Movement; Healthy Volunteer; HV

SUMMARY:
This study will test a spinal cord reflex called reciprocal inhibition before, during, and after learning a motor skill to see if the reflex becomes stronger by learning the movement. People learn new motor skills throughout their lives. At first, performing a new skilled movement such as riding a bicycle takes effort and is clumsy, but with practice, it becomes relatively automatic. The motor cortex (a part of the brain) is very active when a new skilled movement is learned, but becomes less active when the movement is over-learned. This study will determine whether the spinal cord helps coordinate the pattern of activity between groups of muscles once a motor skill is learned.

Healthy volunteers between 21 and 65 years of age may be eligible for this study. Candidates are screened with a medical history and neurological examination.

Participants are divided into two groups. Group 1 has movement training sessions only and Group 2 has both movement training sessions and physiology sessions, as follows:

Movement training sessions

For 15 minutes every weekday, participants practice moving their wrist back and forth to make a cursor on the computer screen follow a target. Activity of the arm muscles is monitored with surface electrodes taped to the skin. The sessions continue until the participant can perform the movement well. Group 1 participants return to the clinic a week after the last session to perform the movement again to see if their skill level has changed. Each session lasts about 20 to 30 minutes.

Physiology sessions

In three separate sessions, the reflex for reciprocal inhibition is measured before and at several times during the movement task. This is done with nerve conduction studies. A probe placed on the skin delivers a low-intensity electrical stimulus. Wires taped to the skin record the nerve impulses. To measure reciprocal inhibition, several dozen stimuli are given to two nerves in combinations. Each session lasts 2 to 3 hours.

DETAILED DESCRIPTION:
Objective:

Once a skilled movement is thoroughly learned, it can be performed relatively automatically. The motor cortex is active when learning a new motor skill, but becomes less activated once the skill has become over-learned. We hypothesize that learning a skilled movement is associated with more efficient use of subcortical motor circuits. Subcortical motor circuits can coordinate features of the intended movement such as the timing and patterns of activation of different muscles. The goal of this study is to determine whether learning a motor skill strengthens spinal interneuron circuits that facilitate the movement. Subjects will learn to perform a movement consisting of alternating wrist movements. The strength of reciprocal inhibition between antagonist muscles will be tested.

Study Population:

22 healthy adult volunteers

Design:

The study has two experiments. Both experiments use a within-subjects design. The purpose of the first experiment is to determine whether learning to accurately perform an alternating wrist flexion and extension movement task is associated with reduced co-contraction of wrist flexor and extensor muscles. Subjects will practice making accurate wrist flexions and extensions to keep a cursor on a target for fifteen-minute sessions every weekday until they are able to obtain 95% accuracy. Activity of the arm muscles will be monitored during the sessions with surface electrodes on the arm muscles. The first experiment will also determine the best training parameters for learning the task. In the second experiment, a second group of subjects will learn the task using the best training parameters. The strength of the reflex for reciprocal inhibition will be measured before, during and after training. Reciprocal inhibition will also be measured after the movement has become highly learned.

Outcome measures:

In the first experiment, the outcome will be the percent of movement time in which co-contraction occurs, as recorded from surface electrodes, while the subject learns to perform the movement to 95% accuracy. In the second experiment, the outcome measure is the strength of spinally mediated reciprocal inhibition, as measured using reflexes.

ELIGIBILITY:
INCLUSION CRITERIA:

Healthy individuals between the ages of 21-65 years who are willing to participate in daily training sessions and physiological studies.

EXCLUSION CRITERIA:

Any history of peripheral nerve injury, cervical radiculopathy, arthritis, tendonitis, or surgery on the wrist.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22
Dates: Start 2004-01; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Pascual-Leone A, Grafman J, Hallett M. Modulation of cortical motor output maps during development of implicit and explicit knowledge. Science. 1994 Mar 4;263(5151):1287-9. doi: 10.1126/science.8122113.
- [Background] Smith ME, McEvoy LK, Gevins A. Neurophysiological indices of strategy development and skill acquisition. Brain Res Cogn Brain Res. 1999 Jan;7(3):389-404. doi: 10.1016/s0926-6410(98)00043-3. PMID 9838200
- [Background] Honda M, Deiber MP, Ibanez V, Pascual-Leone A, Zhuang P, Hallett M. Dynamic cortical involvement in implicit and explicit motor sequence learning. A PET study. Brain. 1998 Nov;121 ( Pt 11):2159-73. doi: 10.1093/brain/121.11.2159. PMID 9827775